CLINICAL TRIAL: NCT04582292
Title: Laryngeal Manifestations of Connective Tissue Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebatullah badry hanafy mahmoud, Principal investigator, Assiut University
Other Study IDs: AssiutUhb
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Connective Tissue Diseases
Keywords: Laryngeal manifestation in connective tissue diseases
MeSH Terms: conditions — Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Connective tissue diseases represent a rather heterogeneous spectrum of overlapping pathologies, which have as a common feature the involvement of multiple organ systems. Though generally uncommon, they represent lifelong conditions, which are often coupled with various immunologic disorders, thus significantly affecting the overall health and quality of life of the affected individual. The classic connective tissue disorders include rheumatoid arthritis ,Juvenile idiopathic arthritis, systemic lupus erythematosus , scleroderma, Sjogren's syndrome, and the mixed connective tissue disease several studies have reported that up to fifty percent of connective tissue diseases' patients are having laryngeal involvement as the sole manifestation of this disease In acute phases, patients may complain of burning, foreign body sensation in the throat, and difficulty in swallowing. In chronic cases the cricoarytenoid joint is usually affected with resultant fixation. The laryngoscopic findings include mucosal edema, myositis of the intrinsic laryngeal muscles, hyperemia, inflammation and swelling of the arytenoids, interarytenoid mucosa, aryepiglottic folds and epiglottis, and impaired mobility or fixation of the cricoarytenoid joint. In the early stage of the disease, the laryngeal examination may be normal

DETAILED DESCRIPTION:
In acute involvement of the cricoarytenoid joints, signs of inflammation such as edema and redness may be present with or without impaired mobility chronic cases where ankylosis of the connective tissue disease cricoarytenoid joint is present, one or both vocal folds may be fixed in the median, paramedian, or lateral positions. Other laryngoscopic findings include the presence of inflammatory masses or rheumatoid nodules in the larynx and pharynx. In 1987, the American Rheumatism Association has included submucosal nodules in the laryngeal tissue in her revised criteria for the classification of Rheumatoid arthritis there was a description of small submucous rheumatoid nodule in the larynx, were later confirmed by multiple studies . Rheumatoid deposits in the form of bamboo nodes which are white- yellow bands in the middle of the membranous portion of the vocal folds had been described Cricoarytenoiditis has been reported to occur in Juvenile rheumatoid arthritis, and sometimes, it may be the first presentation of the disease ,Vocal cord lesions that have been reported in connective tissue diseases diseases include cricoarytenoid arthritis, rheumatoid nodules, and bamboo nodes .

ELIGIBILITY:
Inclusion Criteria:

1. Age: any age group may be included in this study.
2. Gender: both sexes will be included in the study.
3. 'previously established diagnosis of connective tissue diseases:

Exclusion Criteria:

1. history of neurological diseases .
2. previous history of neck radiation
3. presence of any other systemic diseases
4. professional voice users
5. chronic nonspecific laryngitis like laryngeal scleroma,Tuberculous laryngitis
6. presence of laryngeal masses
7. history of neurological diseases .
8. previous history of neck surgery,intubation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cross_sectional study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective measurement of severity of dysphonia connective tissue disease. | Baseline
  Measurement of grades of dysphonia,strain,leakiness,breathiness and irregularity by auditory perceptual assessment using modified GrBAS scale,grades from normal 0 to severe 3
Subjective measurements of patient's assessment of voice severity | Baseline
  Measurement of scores of Arabic voice handicap index
Objective measurement of vocal pitch | Baseline
  Measurement of acoustic analysis (fundamental frequency)
Objective measurement of vocal waveform frequency aperiodicity | Baseline
  Measurement of acoustic analysis (jitter%)
Objective measurement of vocal waveform amplitude aperiodicity | Baseline
  Measurement of acoq1qustic analysis (shimmer%)
Objective measurement of vocal waveform periodicity to aperiodicity ratio | Baseline
  Measurement of acoustic analysis :harmonic to noise ratio (db)

SECONDARY OUTCOMES:
Objective measurements of changes of vocal folds | Baseline
  Measurement of amplitude,symmetry,periodicity,glottal closure and mucosal wave using video_rhino_laryngo_stroboscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: Hebatullah Badry, Bachelor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gaubitz M. Epidemiology of connective tissue disorders. Rheumatology (Oxford). 2006 Oct;45 Suppl 3:iii3-4. doi: 10.1093/rheumatology/kel282. PMID 16987829
- [Background] Silman AJ, Pearson JE. Epidemiology and genetics of rheumatoid arthritis. Arthritis Res. 2002;4 Suppl 3(Suppl 3):S265-72. doi: 10.1186/ar578. Epub 2002 May 9. PMID 12110146
- [Background] Friedman BA. Rheumatoid nodules of the larynx. Arch Otolaryngol. 1975 Jun;101(6):361-3. doi: 10.1001/archotol.1975.00780350025006. PMID 1131102
- [Background] Upile T, Jerjes W, Sipaul F, Singh S, Hopper C, Wright A, Sandison A. Rheumatoid nodule of the thyrohyoid membrane: a case report. J Med Case Rep. 2007 Oct 31;1:123. doi: 10.1186/1752-1947-1-123. PMID 17974016
- [Background] Woo P, Mendelsohn J, Humphrey D. Rheumatoid nodules of the larynx. Otolaryngol Head Neck Surg. 1995 Jul;113(1):147-50. doi: 10.1016/S0194-59989570160-5. PMID 7603711
- [Background] Van der Goten A. Evaluation of the patient with hoarseness. Eur Radiol. 2004 Aug;14(8):1406-15. doi: 10.1007/s00330-004-2272-x. Epub 2004 Apr 14. PMID 15085384
- [Background] Petty RE, Southwood TR, Baum J, Bhettay E, Glass DN, Manners P, Maldonado-Cocco J, Suarez-Almazor M, Orozco-Alcala J, Prieur AM. Revision of the proposed classification criteria for juvenile idiopathic arthritis: Durban, 1997. J Rheumatol. 1998 Oct;25(10):1991-4. No abstract available. PMID 9779856
- [Background] Jacobs JC, Hui RM. Cricoarytenoid arthritis and airway obstruction in juvenile rheumatoid arthritis. Pediatrics. 1977 Feb;59(2):292-4. PMID 834514
- [Background] Hosako-Naito Y, Tayama N, Niimi S, Aotsuka S, Miyaji M, Oka T, Fujinami M, Kitahara N. Diagnosis and physiopathology of laryngeal deposits in autoimmune disease. ORL J Otorhinolaryngol Relat Spec. 1999 May-Jun;61(3):151-7. doi: 10.1159/000027661. PMID 10325555
- [Background] Hilgert E, Toleti B, Kruger K, Nejedlo I. Hoarseness due to bamboo nodes in patients with autoimmune diseases: a review of literature. J Voice. 2008 May;22(3):343-50. doi: 10.1016/j.jvoice.2006.10.009. Epub 2007 Feb 5. PMID 17280816
- [Background] SCARPELLI DG, McCOY FW, SCOTT JK. Acute lupus erythematosus with laryngeal involvement. N Engl J Med. 1959 Oct 1;261:691-4. doi: 10.1056/NEJM195910012611404. No abstract available. PMID 14442250